CLINICAL TRIAL: NCT06742684
Title: Hyperoxemic Oxygen Therapy in Patients With Acute Anterior Myocardial Infarction
Acronym: HOT-AAMI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study could not be started due to a lack of funding for the provision of the medical product to be investigated.
Sponsor: IHF GmbH - Institut für Herzinfarktforschung (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO-001
Record Dates: First submitted 2024-12-13; First posted 2024-12-19 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Myocardial Infarction (MI)
Keywords: AMI; PCI; Hyperoxemic Therapy
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Only PCI (No Intervention): Patients only will receive a PCI according to standard of care
- PCI with following SSO2 Therapy (Experimental): Patient receive a PCI according to standard of care. Additionally patients in this arm will be treated right after the PCI with the SSO2 Therapy
  Interventions: Procedure: PCI with following SSO2 Therapy

INTERVENTIONS:
Procedure: PCI with following SSO2 Therapy — SSO2 Therapy
  Arms: PCI with following SSO2 Therapy

SUMMARY:
The HOT-AAMI study investigates the efficacy of supersaturated oxygen therapy (SSO2) as an adjunct to standard percutaneous coronary intervention (PCI) with stent implantation in patients suffering from acute anterior myocardial infarction (AMI). This is a prospective, open-label, multicenter, two-arm, randomized (1:1) clinical trial conducted in Germany.

Objective:

The primary aim is to assess whether SSO2 therapy reduces the risk of mortality and heart failure progression after PCI compared to PCI alone. Secondary endpoints include cardiac morbidity, quality of life (Kansas City Cardiomyopathy Questionnaire), and adverse events over 12 months.

Study Design:

The trial involves 1,266 patients randomized to receive either the SSO2 therapy post-PCI or PCI alone. Participants must be adults with acute anterior AMI and undergo successful PCI within 6 hours of symptom onset. Recruitment is expected to span 36 months with a follow-up period of 12 months for each participant.

Intervention and Control:

Intervention group: SSO2 therapy delivered intracoronary using hyperoxygenated blood.

Control group: Standard PCI with stent placement without adjunctive therapy.

Primary Endpoint:

The combined outcome of all-cause mortality or unplanned hospital/ambulatory visits for heart failure requiring intravenous diuretics within 12 months post-randomization.

Background and Rationale:

AMI treatment often leaves significant myocardial damage despite successful PCI. Prior studies on SSO2 therapy have demonstrated potential benefits, including reduced infarct size and improved myocardial function, with evidence suggesting reduced heart failure rates and improved long-term survival.

Statistical Power:

The study anticipates a primary endpoint event rate of 16% in the control group, with a hypothesized hazard reduction of 25% in the intervention group. A total of 393 events across 1,266 patients are needed to achieve an 80% power at a 5% significance level.

Safety and Monitoring:

A Data Safety Monitoring Board (DSMB) will oversee the trial. Adverse events will be documented and reported according to protocol guidelines.

Expected Outcomes:

If successful, the study may provide evidence for integrating SSO2 therapy into clinical practice, potentially lowering mortality and morbidity in AMI patients, with implications for both patient care and healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

Inclusion criteria that must be present before PCI:

* Age ≥18 years
* Presence of an acute anterior wall infarction with ST-segment elevation ≥ 1mm in two or more contiguous leads V1 - V4, or newly developed left bundle branch block
* Symptom duration ≤6 hours
* Systemic arterial oxygen partial pressure (pO2) of at least 10.7 kPa or 80 mmHg
* Written informed consent, or procedures following Article 68 MDR Clinical Trials in emergencies

Angiographic Inclusion Criteria:

These criteria are assessed after the study participant has signed the informed consent form and coronary angiography and PCI have been performed.

• Successful PCI of the proximal or middle LAD (left anterior descending artery). Success is defined as a residual stenosis of <50% in all treated culprit lesions with a TIMI flow (Thrombolysis in Myocardial Infarction) of ≥2 in the target vessel.

Exclusion Criteria:

General Exclusion Criteria:

* Previous coronary bypass surgery involving the LAD
* Previous anterior wall infarction with known ischemic cardiomyopathy
* Active bleeding, bleeding diathesis, or a history of coagulopathy (including heparin-induced thrombocytopenia)
* Known intracerebral tumor, aneurysm, arteriovenous malformation, or a history of hemorrhagic stroke
* Known prior organ transplantation or on the waiting list
* Severe mitral regurgitation, ventricular septal defect, ischemic myocardial rupture, or other mechanical complications of acute myocardial infarction
* Acute aortic dissection
* Known severe valvular stenosis or insufficiency, pericardial disease, or non-ischemic cardiomyopathy
* The patient belongs to a particularly vulnerable population or suffers from a significant medical or social condition that, in the investigator's opinion, could impair the patient's ability to participate in the study or comply with follow-up procedures (e.g., alcoholism, dementia, living far from the study site, etc.)
* Current participation in another study involving an investigational product or drug
* Patients who develop any of the following complications in the catheterization lab before completing the PCI procedure: cardiogenic shock (systolic blood pressure: SBP less than 80 mmHg for more than 30 minutes), emergency placement of an intra-aortic balloon pump (IABP), an Impella pump, or ECMO (extracorporeal membrane oxygenation), or cardiopulmonary resuscitation for > 10 minutes.

Angiographic Exclusion Criteria:

• Left main coronary artery stenosis more than 80%.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality or unplanned heart failure hospital admission or unplanned outpatient visit due to heart failure requiring intravenous diuretic therapy | 12 months after the last patient is enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Zeymer, Prof Dr, Principal Investigator — IHF GmbH

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zeymer U, Hassinger F, Bramlage P, Schafer A, Westermann D, Thiele H; HOT-AAMI Investigators. Hyperoxemic oxygen therapy in patients with acute anterior myocardial infarction: HOT-AAMI-design and rationale of a randomized trial. Am Heart J. 2025 Aug;286:35-44. doi: 10.1016/j.ahj.2025.03.013. Epub 2025 Mar 21. PMID 40122364